CLINICAL TRIAL: NCT05894122
Title: Evaluation of Capillary Blood Collection Devices (Mitra® and HemaPEN®) in the Context of Metabolic Diseases and, in Particular, Pediatric Monitoring of Phenylketonuria
Brief Title: Evaluation of Capillary Blood Collection Devices (Mitra® and HemaPEN®)
Acronym: MitrAlanine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC22.0319; 2023-A01180-45 (Other: ID RCB)
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Phenylketonuria; Metabolic Diseases
MeSH Terms: conditions — Phenylketonurias; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood collection on blotters : DM-DIV MITRA® and DM-DIV HemaPEN® for research and Perkin Elmer device for care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DM-DIV MITRA® — Comparison of phenylalanine concentrations in the new device with those in the current device (blotter).
  Other Names: DM-DIV HemaPEN®

SUMMARY:
The aim is to demonstrate a new application for a blood collection device. This device is already widely used in pharmacology. It is not currently used for metabolic diseases.

Its ease of use enables repeated sampling at home. What's more, the device can be sent by post, making it ideally suited to the needs of this cohort of children, whose phenylalanine levels need to be monitored very regularly.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 months to 18 years
* suffering from phenylketonuria or hyperphenylalaninemia
* who have had a capillary and blood test including a phenylalanine assay at CHUGA
* Whose parents or legal guardians are affiliated to the social security system.
* For whom parents or legal guardians have not objected to the MitrAlanine study.

Exclusion Criteria:

* Parents or legal guardians opposed to the MitrAlanine study

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of phenylalanine concentrations | Day 1
  Comparison of phenylalanine concentrations in the new device with those in the current device (blotter).

SECONDARY OUTCOMES:
Ease of use of research device | Day 1
  ease of use of DM-DIV MITRA® and DM-DIV HemaPEN® via a 3 questions-and-answer guide for samplers
sample conformity | Day 1
  Conformity of blood sample on DM-DIV MITRA® and DM-DIV HemaPEN® versus DM-DIV Perkin Elmer
comparison of concentrations of tyrosin | Day 1
  comparison of concentrations of other amino acids (tyrosin) dosed at the same time as phenylalanine
comparison of concentrations of total leucin | Day 1
  comparison of concentrations of other amino acids (total leucin) dosed at the same time as phenylalanine
comparison of concentrations of methionin | Day 1
  comparison of concentrations of other amino acids (methionin) dosed at the same time as phenylalanine

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France